CLINICAL TRIAL: NCT04250103
Title: Developing Innovative Models for Health & Long-term Care Facilities and Technology Services: Prospective Cohort Study for Home Health Care
Brief Title: Home-based Longitudinal Investigation of the Multidisciplinary Team Integrated Care
Acronym: HOLISTIC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Taiwan Society of Home Health Care (Other)
Responsible Party: Principal Investigator, Chao A. Hsiung, Institute of population health sciences, National Health Research Institutes, Taiwan
Other Study IDs: EC1080203
Record Dates: First submitted 2020-01-15; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Health Care Utilization; Caregiver Burnout
Keywords: Home health care; Super-aged society
MeSH Terms: conditions — Patient Acceptance of Health Care; Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient: patients who receive home health care
- caregiver: caregivers who take care of patients with home health care

SUMMARY:
Some research found the effectiveness of implementation of home health care on patients' physical function, quality of life (QoL) and decreased the risk of hospitalization and medical costs. However, little was known about the longitudinal change of comprehensive assessments of physical and mental health, QoL, well-being, and medical resource utilization of patients receiving home health care and their caregivers. Furthermore, the evaluation of advance care planning, palliative care need, and the quality of dying and death were also insufficient among the aforementioned population. Therefore, this cohort study aims to investigate the longitudinal change of health-related outcomes and utilization of resource utilization, and explore their trajectories in two years for patients who receive home health care and their caregivers in Taiwan.

DETAILED DESCRIPTION:
This is a prospective longitudinal cohort study in Taiwan. Data will be collected by trained interviewers at the baseline (T0), 3-month follow-up (T1), 6-month follow-up (T2), 12-month follow-up (T3), 18-month follow-up (T4), and 24-month follow-up (T5). Via home visits, interviewer-administered questionnaires (informed consent, contact/follow-up information, background information, health condition, physical functioning, cognitive function, etc.) will be used. It estimates that the home visit will take up to 2 hours.

The investigators will recruit at least 1200 eligible patients and caregivers (600 dyads) from at least 15 institutions (e.g., home clinics and hospitals) which provide home health care. Trained research assistants will touch based with eligible participants recommended by institution staff and invite them to take part in the study. To ensure the study are achieving the target sample the investigators will examine the distribution of living area and number of participants in each type of home health care unit during recruiting. Moreover, the investigators have estimated an attrition rate of 20% over the study. Higher drop-off rates in certain sub-groups may be problematic, so the investigators will monitor participants' attrition.

In addition, the cohort the investigators enrolled will be linked to their data in Taiwan's National Health Insurance Research Database to analyze the medical resource utilization of participants in our study. The results will show the health status and resource utilization as well as quality of home health care in Taiwan for clinical practices, research and future policy making.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years or older
* Receiving home health care services at least two months
* Either the patient or caregiver can express clearly

Exclusion Criteria:

* Reject to sign the informed consent
* Both the patient and caregiver cannot complete the interview
* Both the patient and caregiver cannot communicate with an interviewer in a familiar language

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with home health care and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from ability to perform activities of daily living (ADL) at two years | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up, 18-month follow-up, 24-month follow-up
  The Barthel Index will be adapted to assess ADL. The total score ranges from 0 to 100, with 100 indicating full independence in doing daily activities.
Change from frailty at two years | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up, 18-month follow-up, 24-month follow-up
  It will be measured by the 9-point Clinical Frailty Scale (CFS). The total score ranges from 1 to 9, with 7 or higher indicating severe frailty, even being terminally ill.
Change from cognitive function/memory at two years | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up, 18-month follow-up, 24-month follow-up
  It will be measured by the Brain Health Test (Chinese version) via testing the orientation to time, immediate and delayed recall of five items, categorical verbal fluency test. The total score ranges from 0 to 16, with higher scores indicating worse cognitive impairment.
Change from percentage of participants with Dementia at two years | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up, 18-month follow-up, 24-month follow-up
  The Functional Assessment Staging Test (FAST) will be adapted to assess an individual's stage of Alzheimer's disease. It includes seven stages from normal aging to sever Dementia.
Change from mean score of depression at two years | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up, 18-month follow-up, 24-month follow-up
  It will be measured by the 5-item Geriatric Depression Scale (GDS). The total score ranges from 0 to 5, with higher scores indicating more depression.
Change from neuropsychiatric status at two years | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up, 18-month follow-up, 24-month follow-up
  It will be measured by the Neuropsychiatric Inventory. The 10 sub-domains of behavioral functioning are examined, including delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, and aberrant motor activity syndrome.
Change from quality of life (QOL) at two years | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up, 18-month follow-up, 24-month follow-up
  We will adapt the Quality of Life in Alzheimer's Disease (QOL-AD) scale for patients with cognitive impairment, and Quality of Life Survey for Home Care (QOL-HC) scale for those without cognitive impairment. The total score of QOL-AD ranges from 13 to 52, with higher values indicating a higher QoL. The total score of QOL-HC ranges from 0 to 8, with higher values indicating a higher QoL.
Change from mental wellbeing at two years | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up, 18-month follow-up, 24-month follow-up
  It will be measured by the World Health Organization- Five Well-Being Index (WHO-5). The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life.
Shared decision making (SDM) | Two years
  It will be measured by the Decision-making Participation Self-Efficacy Scale (DEPS). The total score ranges from 5 to 25, with higher scores indicating higher self-efficacy.
Advance Care Planning (ACP) | Two years
  It will be measured by the 4-question version of UCSF-ACP with the Process Measures (knowledge, contemplation, self-efficacy, and readiness, 5-point Likert scales) and Action Measures (yes/no whether an ACP behavior is completed).
Change from Nutrition status at two years | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up, 18-month follow-up, 24-month follow-up
  It will include the Mini Nutritional Assessment (MNA). The total score of MNA ranges from 0-14, with more than 11 indicating normal nutrition status.
Change from risk for pressure injury at two years | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up, 18-month follow-up, 24-month follow-up
  It will be measured by the sale of Braden Scale for Predicting Pressure Sore Risk. The scale is composed of six subscales that reflect sensory perception, skin moisture, activity, mobility, friction and shear, and nutritional status. The total score ranges from 6 to 23, with higher scores indicating lower risk for forming pressure sores.
Needs assessment for supportive & palliative care | Two years
  It will be measured by the Supportive & Palliative Care Indicators Tool (SPICT). Following the guideline, the Chinese version will be developed before the cohort study starts.
Change from medical resource utilization at two years | Baseline, 3-month follow-up, 12-month follow-up, 24-month follow-up
  Assessments include medical costs and out-of-pocket costs regarding utilization of medical resource and home health care. The used scales are developed by our research team.
Change from caregiving burden at two years | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up, 18-month follow-up, 24-month follow-up
  It will be measured by the revised version of Zarit Burden interview containing 22 items, with higher scores indicating greater burden.
Change from number of used chronic disease drug at two years | Baseline, 3-month follow-up, 6-month follow-up, 12-month follow-up, 18-month follow-up, 24-month follow-up
  It will be measured by two items which are developed by our research team. Based on patients' prescriptions, they will be required to answer the number of chronic disease drug they used and these drugs' information, including the names, administrations and dosages.

CONTACTS AND LOCATIONS:
Overall Officials: Chao A. Hsiung, PhD, Study Director — National Health Research Institutes, Taiwan; Sang-Ju Yu, MD, Principal Investigator — Taiwan Society of Home Health Care and Home Clinic Dulan; Ping-Jen Chen, MD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Chao A. Hsiung, Zhunan, Miaoli County, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin CP, Liao JY, Huang CH, Cheng SY, Tseng WZ, Mori M, Chang HC, Li CM, Sun WJ, Wu CY, Chiou HY, Yu SJ, Hsiung CA, Chen PJ; HOLISTIC Investigators. Association Between Current Medical Decision-Making Participation Self-Efficacy and Advance Care Planning Engagement Among Older Adults: Baseline Findings from a Nationwide Longitudinal Cohort Study. J Palliat Med. 2025 Jan;28(1):50-58. doi: 10.1089/jpm.2024.0106. Epub 2024 Dec 5. PMID 39636682
- [Derived] Lai YC, Tsai KT, Ho CH, Liao JY, Tseng WZ, Petersen I, Wang YC, Chen YH, Chiou HY, Hsiung CA, Yu SJ, Sampson EL, Chen PJ. Mortality rate and its determinants among people with dementia receiving home healthcare: a nationwide cohort study. Intern Emerg Med. 2023 Oct;18(7):2121-2130. doi: 10.1007/s11739-023-03319-3. Epub 2023 May 30. PMID 37253992
- [Derived] Liao JY, Chen PJ, Wu YL, Cheng CH, Yu SJ, Huang CH, Li CM, Wang YW, Zhang KP, Liu IT, Umegaki H, Hamano J, Mori M, Petersen I, Sampson EL, Hsiung CA. HOme-based Longitudinal Investigation of the multidiSciplinary Team Integrated Care (HOLISTIC): protocol of a prospective nationwide cohort study. BMC Geriatr. 2020 Nov 27;20(1):511. doi: 10.1186/s12877-020-01920-1. PMID 33246407